CLINICAL TRIAL: NCT00932126
Title: Phase 1, Open Label, Dose-Escalation, Safety, Pharmacokinetic And Pharmacodynamic Study Of Single Agent PF-03758309, An Oral PAK4 Inhibitor, In Patients With Advanced Solid Tumors
Brief Title: This Is The First Study Using Escalating Doses Of PF-03758309, An Oral Compound, In Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1301001
Record Dates: First submitted 2009-06-30; First posted 2009-07-03 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Advanced Solid Tumors
Keywords: Phase 1 dose escalation dose finding pharmacokinetic and pharmacodynamic study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-03758309

INTERVENTIONS:
Drug: PF-03758309 — Oral PF-03758309 will be administered in capsules (once or twice daily) until toxicity, progressive disease, or patient refusal to continue on therapy. The starting dose is 1 mg once daily.

SUMMARY:
This is the first study using PF-03758309, an oral compound, in patients with advanced solid tumors. In this study different doses of PF-03758309 will be administered to different groups of patients. The study will assess the compound's safety, the blood levels of PF-03758309 during the treatment and the effect of the compound on the tumor cells.

DETAILED DESCRIPTION:
The study was prematurely terminated on 26Jul2011 due to the undesirable PK characteristics of PF-03758309 and the lack of an observed dose-response relationship. There were no safety concerns that contributed to the study termination.

ELIGIBILITY:
Inclusion Criteria:

* Advanced/metastatic solid tumor that is resistant to standard therapy or for which no standard therapy is available.
* ECOG (Eastern Cooperative Oncology Group) Performance Status (PS) must be 0 or 1.
* Adequate bone marrow, liver and kidney function.

Exclusion Criteria:

* Patients with known brain metastases.
* Previous high dose chemotherapy requiring stem cell rescue.
* Prior irradiation to >25% of the bone marrow.
* Active bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV).
* Current active treatment in another clinical study.
* Pregnancy or breast feeding.
* Active inflammatory gastrointestinal disease, chronic diarrhea (unless related to underlying malignancy or prior related treatment) or history of abdominal fistula, gastrointestinal perforation, peptic ulcer disease, or intra-abdominal abscess within 6 months prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (2):
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Aurora, Colorado
- Pfizer Investigational Site, East Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Mpilla GB, Uddin MH, Al-Hallak MN, Aboukameel A, Li Y, Kim SH, Beydoun R, Dyson G, Baloglu E, Senapedis WT, Landesman Y, Wagner KU, Viola NT, El-Rayes BF, Philip PA, Mohammad RM, Azmi AS. PAK4-NAMPT Dual Inhibition Sensitizes Pancreatic Neuroendocrine Tumors to Everolimus. Mol Cancer Ther. 2021 Oct;20(10):1836-1845. doi: 10.1158/1535-7163.MCT-20-1105. Epub 2021 Jul 12. PMID 34253597
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1301001

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-03758309, 1 Milligram (mg) Once Daily (QD): PF-03758309 1 mg administered orally once daily
- PF-03758309, 1 mg Twice Daily (BID): PF-03758309 1 mg administered orally twice daily
- PF-03758309, 2 mg BID: PF-03758309 2 mg administered orally twice daily
- PF-03758309, 10 mg BID: PF-03758309 10 mg administered orally twice daily
- PF-03758309, 20 mg BID: PF-03758309 20 mg administered orally twice daily
- PF-03758309, 40 mg BID: PF-03758309 40 mg administered orally twice daily
- PF-03758309, 50 mg BID: PF-03758309 50 mg administered orally twice daily
- PF-03758309, 60 mg BID: PF-03758309 60 mg administered orally twice dailly
Period: Overall Study
Arm/Group | PF-03758309, 1 Milligram (mg) Once Daily (QD) | PF-03758309, 1 mg Twice Daily (BID) | PF-03758309, 2 mg BID | PF-03758309, 10 mg BID | PF-03758309, 20 mg BID | PF-03758309, 40 mg BID | PF-03758309, 50 mg BID | PF-03758309, 60 mg BID
Started | 3 | 3 | 3 | 3 | 5 | 3 | 5 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 5 | 3 | 5 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Objective progression or relapse | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 5
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- PF-03758309: Participants who received: 1 mg QD, 1 mg BID, 2 mg BID, 10 mg BID, 20 mg BID, 40 mg BID, 50 mg BID and 60 mg BID
Arm/Group | PF-03758309
Number analyzed (Participants) | 35
Age, Customized [Number; unit: participants]
  <18 years | 0
  18 - 44 years | 6
  45 - 64 years | 15
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cycle 1 Dose-limiting Toxicities (DLT)
Description: DLT includes: Grade (GR) 4 neutropenia (NP) that persisted for >7 consecutive days; Febrile NP; GR3 NP infection; GR4 thrombocytopenia (TP); GR3 TP with bleeding; Any other GR>=3 toxicity not classified under Common Terminology Criteria for Adverse Events (CTCAE) blood or bone marrow (exception of nausea, vomiting, or diarrhea in subjects who received optimal treatment with antiemetics or anti-diarrheals); Failure to recover to an adequate condition to recommence study treatment after a 2-week delay; Failure to receive >= 80% of planned PF-03758309 dose due to study drug related toxicity
Time Frame: Baseline (up to 30 days prior to first study drug administration) till 28 days after the last treatment administration (end of Cycle 1 [28 days])
Population: Safety analysis set: All participants enrolled in the study that received at least 1 dose of PF-03758309 (including the lead in dose).
Measure: Number; unit: participants
Groups:
- PF-03758309, 1 mg QD: PF-03758309 1 mg administered orally once daily
- PF-03758309, 1 mg BID: PF-03758309 1 mg administered orally twice daily
- PF-03758309, 60 mg BID: PF-03758309 60 mg administered orally twice daily
Arm/Group | PF-03758309, 1 mg QD | PF-03758309, 1 mg BID | PF-03758309, 2 mg BID | PF-03758309, 10 mg BID | PF-03758309, 20 mg BID | PF-03758309, 40 mg BID | PF-03758309, 50 mg BID | PF-03758309, 60 mg BID
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 3 | 5 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

2. Secondary Outcome: Number of Participants With Objective Response
Description: Number of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as ≥30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study ≥4 weeks after initial documentation of response.
Time Frame: Baseline until the date of first documented progression or discontinuation from the study due to any cause, assessed every 2 months until when the last participant was discontinued due to disease progression in Month 27 of the study
Population: Per protocol analysis set: all participants who have received a minimum of 1 cycle of study treatment (at least 80% of planned dose), had baseline assessments and at least 1 on-study tumor assessment were considered evaluable for response.
Measure: Number; unit: participants
Groups:
- PF-03758309, 10 mg BID: PF-03758309, 10 mg BID PF-03758309 10 mg administered orally twice daily
Arm/Group | PF-03758309, 1 mg QD | PF-03758309, 1 mg BID | PF-03758309, 2 mg BID | PF-03758309, 10 mg BID | PF-03758309, 20 mg BID | PF-03758309, 40 mg BID | PF-03758309, 50 mg BID | PF-03758309, 60 mg BID
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 3 | 5 | 10
participants
  confirmed complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  confirmed partial response (PR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Time in weeks from start of study treatment to first documentation of objective tumor progression or death due to cancer, whichever comes first. TTP was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD])
Time Frame: as for outcome 2
Population: Data not analyzed due to early termination of the study.
Groups:
- PF-03758309: Participants who received: 1 mg QD, 1 mg BID, 2 mg BID, 10 mg BID, 20 mg BID, 40 mg BID, 50 mg BID, and 60 mg BID
Arm/Group | PF-03758309
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 2
Population: Data not analyzed due to early termination of the study.
Arm/Group | PF-03758309
Number analyzed (Participants) | 0

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: predose, 0.5, 1, 2, 3, 5, 8, 10, 24 and 48 hours post dose, on Cycle 1 Day 8 and Cycle 2-4 Day 1 at pre-dose and 2 hours post morning dose, and on Cycle 1 Day 15 at predose, 0.5, 1, 2, 3, 5, 8 and 10 hours post morning dose
Population: Data not analyzed due to early termination of the study.
Arm/Group | PF-03758309
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 5
Population: Data not analyzed due to early termination of the study.
Arm/Group | PF-03758309
Number analyzed (Participants) | 0

7. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: as for outcome 5
Population: Data not analyzed due to early termination of the study.
Arm/Group | PF-03758309
Number analyzed (Participants) | 0

8. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to 12 Hours Post Morning Dose [AUC(0-12)]
Time Frame: pre-dose and 12 hours post morning dose
Population: Data not analyzed due to early termination of the study.
Arm/Group | PF-03758309
Number analyzed (Participants) | 0

9. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin)
Time Frame: predose, 0.5, 1, 2, 3, 5, 8, 10, 24 and 48 hours post dose, and on Cycle 1 Day 15 at predose, 0.5, 1, 2, 3, 5, 8 and 10 hours post morning dose
Population: Data not analyzed due to early termination of the study.
Arm/Group | PF-03758309
Number analyzed (Participants) | 0

10. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau)
Time Frame: as for outcome 9
Population: Data not analyzed due to early termination of the study.
Arm/Group | PF-03758309
Number analyzed (Participants) | 0

11. Secondary Outcome: PAK (p21 Activated Kinase)-Related Pathway Molecule Expression Modulation by PF-03758309 in Tumor and Surrogate Tissue
Time Frame: Screening, 0, 2, 4, and 72 hours post dose Cycle 2 Day 8. A 6th sample of hair follicle could be requested at 6 or 8 hours post-dose if necessary. For fresh tumor tissue, baseline and between Day 8 and 22 of Cycle 1 in participants with accessible tumors
Population: Data not analyzed due to early study termination.
Arm/Group | PF-03758309
Number analyzed (Participants) | 0

12. Secondary Outcome: Baseline Tumor Expression of PAK-related Pathway Molecules and Other Known Biomarkers
Time Frame: Baseline
Population: Data not analyzed due to early study termination.
Arm/Group | PF-03758309
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- PF-03758309, 1 mg QD: PF-03758309, 1 mg administered orally once daily
Arm/Group | PF-03758309, 1 mg QD | PF-03758309, 1 mg BID | PF-03758309, 2 mg BID | PF-03758309, 10 mg BID | PF-03758309, 20 mg BID | PF-03758309, 40 mg BID | PF-03758309, 50 mg BID | PF-03758309, 60 mg BID
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 1/5 | 0/3 | 1/5 | 2/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 5/5 | 3/3 | 5/5 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03758309, 1 mg QD (N=3) | PF-03758309, 1 mg BID (N=3) | PF-03758309, 2 mg BID (N=3) | PF-03758309, 10 mg BID (N=3) | PF-03758309, 20 mg BID (N=5) | PF-03758309, 40 mg BID (N=3) | PF-03758309, 50 mg BID (N=5) | PF-03758309, 60 mg BID (N=10)
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disease Progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03758309, 1 mg QD (N=3) | PF-03758309, 1 mg BID (N=3) | PF-03758309, 2 mg BID (N=3) | PF-03758309, 10 mg BID (N=3) | PF-03758309, 20 mg BID (N=5) | PF-03758309, 40 mg BID (N=3) | PF-03758309, 50 mg BID (N=5) | PF-03758309, 60 mg BID (N=10)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 5 | 8
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Defaecation urgency0 (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 3 | 3 | 6
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 8
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 0 | 2 | 2 | 2 | 3 | 3 | 3 | 4
Influenza like illness (General disorders) | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 2 | 2 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was closed due to pharmacokinetic (PK) issues observed from initial PK data. Individual plasma concentration versus time were listed but final PK analysis and pharmacodynamic analyses were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.